CLINICAL TRIAL: NCT02052037
Title: Egg Ingestion in Adults With Type 2 Diabetes: Effects on Glycemic Control, Anthropometry, Diet Quality and Cardiometabolic Status A Randomized, Controlled, Crossover Trial
Brief Title: Egg Ingestion in Adults With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Griffin Hospital (Other)
Collaborators: American Egg Board (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2013-05
Record Dates: First submitted 2014-01-29; First posted 2014-01-31 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Egg; Glycemic Control; Insulin sensitivity; Diet quality
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Egg inclusion (Experimental): Participants will meet with a registered dietitian and receive instructions for including 2 eggs per day (10 to 14 eggs/week) in their meal plan, while preserving an isocaloric condition relative to the egg exclusion phase. The study dietitian will provide individualized guidance to participants on how to make room for eggs in their diet, while giving them latitude in determining how to adjust for the extra calories from the eggs, to better approximate real-world conditions.
  Interventions: Dietary Supplement: Egg inclusion
- Egg exclusion (Experimental): Participants will meet with the dietitian and receive relevant meal planning guidance and instructions to avoid eggs and specific egg-containing products.
  During both intervention phases, study participants will be advised to eat to their usual state of fullness, and dietary monitoring and weighing will be conducted to ensure that an isocaloric condition is maintained.
  Interventions: Dietary Supplement: Egg exclusion

INTERVENTIONS:
Dietary Supplement: Egg inclusion — Participants will meet with a registered dietitian and receive instructions for including 2 eggs per day (10 to 14 eggs/week)in their meal plan, while preserving an isocaloric condition relative to the egg exclusion phase. The study dietitian will provide individualized guidance to participants on how to make room for eggs in their diet, while giving them latitude in determining how to adjust for the extra calories from the eggs, to better approximate real-world conditions. Treatment phase will last for 12 weeks.
  Arms: Egg inclusion
Dietary Supplement: Egg exclusion — Participants will meet with the dietitian and receive relevant meal planning guidance and instructions to avoid eggs and specific egg-containing products.
  During both intervention phases, study participants will be advised to eat to their usual state of fullness, and dietary monitoring and weighing will be conducted to ensure that an isocaloric condition is maintained. Treatment phase will last for 12 weeks.
  Arms: Egg exclusion

SUMMARY:
We propose a prospective, randomized, single-blind controlled crossover study to assess the effects of daily egg inclusion versus egg exclusion, on glycemic control, anthropometric measures, and overall diet quality in adults with Type 2 diabetes.

DETAILED DESCRIPTION:
Hypothesis Inclusion of eggs in the diets of individuals with Type 2 diabetes mellitus will improve glycemic control, anthropometric measures and overall diet quality.

Restriction of dietary cholesterol, and thus the avoidance or restriction of egg intake, is routinely recommended to patients at increased risk for CVD, including those with diabetes. However, the relative importance of dietary cholesterol to serum lipids and the role of egg ingestion in cardiovascular risk are increasingly suspect. Further, the exclusion of eggs from the diet may lead to increased consumption of high-glycemic carbohydrate foods of particular potential harm to individuals with diabetes. The examination of how food-specific recommendations translate into effects on other food choices and overall diet quality, and in turn health effects, is a neglected area of research.

Eggs provide a complete profile of amino acids and an array of micronutrients, and are low in total fat. Although epidemiological and clinical studies largely suggest a lack of association between egg intake and harmful effects, the evidence is somewhat more ambiguous with regard to glycemic control for diabetes, or the risk for CVD among individuals with diabetes. Our own prior work shows no adverse effects of egg ingestion in healthy adults, hyperlipidemic adults, or adults with established coronary artery disease. As a satiating and protein-rich food, eggs have potential to foster calorie and weight control, and to reduce the dietary glycemic load, offering potential advantages in Type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* males age greater than 35 years;
* post-menopausal females not currently on hormone replacement therapy;
* non-smokers;
* clinical diagnosis of Type 2 diabetes mellitus for at least 1 year but no more than 5 years;
* 6.5% ≤ HbA1c ≤8.0% (5) BMI between 25 and 40 kg/m².

Exclusion Criteria:

* failure to meet inclusion criteria;
* anticipated inability to complete study protocol for any reason;
* current eating disorder;
* use of antihyperglycemic, lipid-lowering or antihypertensive medications unless stable on medication for at least 3 months;
* use of glucocorticoids, antineoplastic agents, psychoactive agents, or nutraceuticals;
* regular use of fiber supplements;
* restricted diets (i.e., vegetarian, vegan, gluten free);
* known allergy to eggs.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Glycemic Index | 12-weeks
  Glycated hemoglobin A1c (HbA1c) will be used to measure the average plasma glucose concentration.

SECONDARY OUTCOMES:
Fasting glucose and insulin | 12-weeks
  Glucose and insulin will be measured at each time point. Participants will be asked to fast at least 8 hours before glucose and insulin measurement. Homeostasis Model Assessment (HOMA-IR) values will be calculated from fasting serum glucose and serum insulin levels using HOMA calculator version 2.2.1 to gauge the degree of insulin resistance.
Body Composition | 12- weeks
  Body composition will be measured using bioelectrical impedance analysis, which uses the resistance of electrical flow through the body to estimate body fat. The Tanita SC-240 Body Composition Analyzer will be used to measure body composition. The SC-240 Body Composition Analyzer measures weight and calculates body fat% and total body water% in addition to BMI.
Body Weight | 12- weeks
  Body weight will be measured during each visit. It will be measured to the nearest 0.5 pound using a balance-type medical scale. Subjects will be measured in the morning (fasting), unclothed with the exception of undergarments.
Waist Circumference | 12-weeks
  Waist circumference will be measured using the U.S. government standard protocol. It will be measured around the narrowest point between ribs and hips when viewed from the front after exhaling.
Diet Quality | Baseline, 6-weeks, 12-weeks
  To help the study team track any variation in dietary pattern over the course of the study, all participants will be asked at two time points to provide information on the foods and beverages that they consumed during a 3-day period. For each 3-day period, participants will complete three 24-hour recalls using a web-based Automated Self-Administered 24-Hour Recall (ASA24) (available from the National Cancer Institute at http://riskfactor.cancer.gov/tools/instruments/asa24/) which will guide them through the process of completing the recall data. Diet quality will be assessed using the Alternative Healthy Eating Index (AHEI). 3-day food period data will be collected at baseline, 6 weeks and 12 weeks.
Physical Activity | 12-weeks
  Physical activity will be determined by the Seven-Day Physical Activity Recall [PAR]. The PAR is one of the most widely used physical activity assessments in exercise science and epidemiological research. The popularity of this measure stems largely from its versatility and relative ease of use for research applications. The PAR provides detail regarding the duration, intensity, and volume (energy expenditure) of physical activity and can therefore be used for a variety of applications. Because it utilizes a one-week time frame, the data from the PAR is often considered representative of typical activity patterns. While it requires considerable cognitive effort by the participants, the interviewer administered version can be completed in a reasonable amount of time (~20 minutes). Variation in physical activity level will be controlled in our multivariable regression models.

CONTACTS AND LOCATIONS:
Overall Officials: David L. Katz, MPH,MD, Principal Investigator — Yale-Griffin Prevention Research Center; Valentine Y. Njike, MPH,MD, Principal Investigator — Yale-Griffin Prevention Research Center
Locations (1):
- Yale-Griffin Prevention Research Center, Derby, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Njike VY, Annam R, Costales VC, Yarandi N, Katz DL. Which foods are displaced in the diets of adults with type 2 diabetes with the inclusion of eggs in their diets? A randomized, controlled, crossover trial. BMJ Open Diabetes Res Care. 2017 Jul 13;5(1):e000411. doi: 10.1136/bmjdrc-2017-000411. eCollection 2017. PMID 28761662
- [Derived] Njike VY, Ayettey RG, Rajebi H, Treu JA, Katz DL. Egg ingestion in adults with type 2 diabetes: effects on glycemic control, anthropometry, and diet quality-a randomized, controlled, crossover trial. BMJ Open Diabetes Res Care. 2016 Dec 22;4(1):e000281. doi: 10.1136/bmjdrc-2016-000281. eCollection 2016. PMID 28074139